CLINICAL TRIAL: NCT04391192
Title: Virtual Overdose Response
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor determined that it must be terminated
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); AHS Addiction and Mental Health Strategic Clinical Network (Unknown); TELUS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AMH-SCN-05
Record Dates: First submitted 2020-04-28; First posted 2020-05-18 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Drug Overdose
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Intervention Model Description: Feasibility of using a phone line to provide overdose response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): All participants will be given the phone number and encouraged to call any time they plan to use substances alone
  Interventions: Behavioral: Virtual Overdose Response

INTERVENTIONS:
Behavioral: Virtual Overdose Response — All participants will be provided the phone number and encouraged to call when they use alone.

SUMMARY:
To help prevent deaths in populations that cannot or will not access physical safer consumption services in Alberta, which may disproportionately include women and those who are not able to self-inject (Potier et al., 2014) the investigators propose to provide virtual (phone-based) supervised consumption services, staffed by people with lived experience.

DETAILED DESCRIPTION:
Designed as a small open label clinical study to demonstrate proof of concept which will follow CONSORT guidelines, the investigators aim to recruit approximately 15 people who are currently using illicit substances and who currently use opioids (illicit or prescription - non-medically). The sample size of 15 balances pragmatic issues (difficulty in recruiting people who are actively using illicit substances) and the need to have a good sample of the population. These participants will be interviewed by the research coordinator in person prior to intervention initiation to determine baseline use; history of overdose; and current harm reduction activities (see appendix). They will then be asked to call the intervention number if they are going to be using alone (see appendix for call flow).

Each time a participant dials the number, the operator will gather (as part of the intervention) the address the participant is at, their name/pseudonym and a phone number that can be used as a call back number in case the call is disconnected. The phone line operator will then ask a) what they planned on using, b) the method of use, c) if the participant is using safe sterile supplies (and provide information on where they can get new supplies in their community), and d) if they have a naloxone kit (overdose reversal kit) available. They will then inform the participant that they will be checking in on them every 5 - 10 minutes and if they do not respond, they will call emergency medical services for them.

If the participant responds to each verbal prompt (calling their name) over a minimum of 30 minutes, the operator will let them know that they are disconnecting the call. The operator will offer to connect the participant to other health services, such as the location of new supplies, social services, addiction treatment and opioid agonist therapy. If the participant fails to respond to a prompt (or the call is disconnected and is not able to be reconnected), the operator will contact the dispatch supervisor and the process for emergency services dispatch will be initiated.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent - able to speak and understand English and over 18 years of age
* Admit to using opioids non-medically: using illicit opioids; using prescription opioids without a current prescription; using doses greater than those prescribed; using opioids recreationally
* Have access to a phone line in the location they primarily use opioids: this can be a land line or a cell phone
* Resident of Calgary

Exclusion Criteria:

* Unable to give informed consent - unable to understand English, under 18 years of age or otherwise not legally able
* Do not knowingly use opioids non-medically
* No access to a phone
* Live outside of Calgary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Usage | 3 months
  Number of times participants call the phone line

SECONDARY OUTCOMES:
EMS response time | 3 months
  Amount of time from calling 911 to EMS arriving on scene
EMS dispatch outcome | 3 months
  qualitative description of dispatch outcome

OTHER OUTCOMES:
Length of calls | 3 months
  overall time required for a single call to the service
Proportion of calls for which EMS is dispatched | 3 months
  quantitative analysis of the number of times the operator calls 911 for a participant
Timing of calls | 3 months
  Analysis of what time of day most calls come in to the service
Health care usage | 3 months
  analysis of overall health system usage (based on administrative data) by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Rittenbach, PhD, Principal Investigator — Alberta Health services
Locations (1):
- Undetermined, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD

REFERENCES:
- [Derived] Bristowe SK, Ghosh SM, Trew M; Canadian Mental Health Association - Calgary Region; Rittenbach K. Virtual Overdose Response for People Who Use Opioids Alone: Protocol for a Feasibility and Clinical Trial Study. JMIR Res Protoc. 2021 May 12;10(5):e20183. doi: 10.2196/20183. PMID 33978598